CLINICAL TRIAL: NCT05142449
Title: Effect of Systemic Antibiotic Therapy on Postoperative Complications in Patients Undergoing Wisdom Teeth Removal Surgery. A Double-blind, Randomised, Placebo-controlled Trial
Brief Title: Effect of Systemic Antibiotic Therapy on Postoperative Complications in Patients Undergoing Wisdom Teeth Removal Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AMOXI
Record Dates: First submitted 2021-11-24; First posted 2021-12-02 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Third Molar Extraction Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amoxilan (Experimental): Patients receive 8 capsules Amoxilan perioperatively and for the next 3 days 6 capsules per day.
  Interventions: Drug: Amoxilan
- Placebo (Placebo Comparator): Patients receive 8 capsules Placebo perioperatively and for the next 3 days 6 capsules per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxilan — Patients receive 8 capsules Amoxilan perioperatively and for the next 3 days 6 capsules per day
  Arms: Amoxilan
Other: Placebo — Patients receive 8 capsules placebo perioperatively and for the next 3 days 6 capsules per day
  Arms: Placebo

SUMMARY:
59 medically healthy patients, who are scheduled for third molar extraction surgery and give informed consent for the trial, are operated using a split-mouth technique.

One group of patients will be assigned to the test group (Amoxilan) for the first surgery and to the control group (placebo) for the second surgery, and vice versa, according to randomisation.

Patients receive 8 capsules Amoxilan or placebo (according to randomisation) perioperatively, and 6 capsules Amoxilan/placebo per day for 3 days postoperativeley.

ELIGIBILITY:
Inclusion Criteria:

* Symptom-free, bilaterally located third molars
* Medically healthy patient ≥ 16 years
* No allergies/intolerances against the investigational product/placebo
* Informed consent

Exclusion Criteria:

* General contraindications to wisdom tooth extraction surgery
* (Former) heavy smoking
* Use of antibiotics within the last three months or patients requiring antibiotic treatment prior to surgery
* (Planned) Pregnancy/lactating

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Mouth opening restrictions: Change of interincisal distance | preoperatively as well as on the 1st and 7th postoperative day
  Interincisal distance, with maximum mouth opening, is measured with a ruler.

SECONDARY OUTCOMES:
Change of swelling | preoperatively as well as on the 1st and 7th postoperative day
  Swelling in the cheek area will be determined using a tape measure and 3D photographs.
Change of Visual Analogue Scale (VAS): Bleeding | day of surgery, and on day 1, 2, 3, 4, 5, 6, 7 after surgery
  Patients indicate bleeding symptoms on a VAS scale, ranging from 0-10, whereas higher values indicate a worse outcome
Change of Visual Analogue Scale (VAS): Swelling | day of surgery, and on day 1, 2, 3, 4, 5, 6, 7 after surgery
  Patients indicate swelling on a VAS scale, ranging from 0-10, whereas higher values indicate a worse outcome
Change of Visual Analogue Scale (VAS): Pain | day of surgery, and on day 1, 2, 3, 4, 5, 6, 7 after surgery
  Patients indicate pain on a VAS scale, ranging from 0-10, whereas higher values indicate a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Universität Graz, Klin. Abteilung für Orale Chirurgie und Kieferorthopädie, Graz, Austria